CLINICAL TRIAL: NCT02515773
Title: MOBILITY- Metformin for Overweight & OBese ChILdren and Adolescents With BIpolar Spectrum Disorders Treated With Second-Generation AntipsYchotics
Brief Title: Metformin for Overweight & OBese ChILdren and Adolescents With BDS Treated With SGAs
Acronym: MOBILITY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melissa Delbello (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Melissa Delbello, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DelBello PCORI
Record Dates: First submitted 2015-07-31; First posted 2015-08-05 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MET and LIFE (Experimental): Participants randomized to this group will receive both Metformin and lifestyle intervention.Participants randomized to treatment with MET will start at a dose of 500 mg orally at night and slowly titrated in 2-week intervals to ensure that each patient achieves maximum insulin-sensitizing effects of the drug while minimizing the chance of side effects. Investigators will also recommend that MET be taken with food to minimize side effects. If a participant's BMI percentile <5% (=underweight) his/her treatment with MET will be discontinued. Although the risk of low vitamin B12 while taking MET is associated with age > 50 years and having type II diabetes, Investigator will monitor B12 levels and a CBC throughout study participation.
  Interventions: Drug: Metformin; Behavioral: healthy lifestyle intervention (LIFE)
- Healthy lifestyle intervention (LIFE) (Experimental): Participants randomized to this group will receive just lifestyle intervention alone.This healthy lifestyle intervention (LIFE) consists of counseling participants and families regarding a healthy eating plan, physical activity and sedentary activities. Prior to study initiation, clinical site staff will participate in a live (or taped) training session from a dietician to lean to administer LIFE. A trained site staff member (e.g. medical assistant or case manager) will meet with participants and their families for a 15-20 minute session at baseline that will focus on nutritional issues using the Traffic Light Plan (TLP).
  Interventions: Behavioral: healthy lifestyle intervention (LIFE)

INTERVENTIONS:
Drug: Metformin — Metformin - to achieves maximum insulin-sensitizing effects
  Other Names: GLUCOPHAGE
  Arms: MET and LIFE
Behavioral: healthy lifestyle intervention (LIFE) — Healthy Life style intervention
  Other Names: LIFE

SUMMARY:
A prospective, large, pragmatic, randomized trial to study the impact of METFORMIN and healthy lifestyle intervention (LIFE) vs. LIFE alone on patient-centered outcomes of body weight, SGA-adherence and satisfaction, psychiatric symptom burden (e.g. mood/anxiety), and Quality of Life.

DETAILED DESCRIPTION:
The investigators propose to recruit 1800 overweight/obese youth with Bipolar Spectrum Disorder (BSD) who are prescribed second generation anti psychotics (SGAs) from at least 24 public and private mental health practices in the Greater Cincinnati and New York City regions, (approximately 900 each from ~12 Cincinnati region and ~12 Long Island/New York mental health treatment sites) to participate in the proposed patient-centered large pragmatic trial examining the effectiveness of MET and LIFE vs. LIFE alone. Patients will be eligible if they are ages 8-17 years old, inclusive, overweight or obese (BMI > 85%), continuing or starting treatment with at least one SGA (i.e., olanzapine, clozapine, risperidone, quetiapine, aripiprazole, ziprasidone, iloperidone, lurasidone, paliperidone, or asenapine) and have a clinical diagnosis of BSD (bipolar I or II disorder, cyclothymia, or bipolar or mood disorder not otherwise specified [or by Diagnostic and Statistical Manual of Mental Disorders V (DSM-5), other specified bipolar or mood disorder). The enrollment rate will be 2-3 patients/month/site for a recruitment time of 30 months.

ELIGIBILITY:
Inclusion Criteria

1. Inpatient or outpatient age 8-19 years inclusive; participants must live with a parent, guardian, or caregiver;
2. Fluent in English;
3. Diagnosed or told by a clinician that they have any of the following bipolar spectrum disorders (BSD): bipolar I, bipolar II, unspecified bipolar and related disorders, Disruptive Mood Dysregulation Disorder (DMDD), cyclothymic disorder, other specified bipolar and related disorders, as well as mood disorder not otherwise specified (if diagnosed in the past as per DSM-IV);
4. Body mass index >85%ile for age and sex by standard growth charts;
5. Received a new or ongoing prescription for at least one SGA (i.e., olanzapine, clozapine, risperidone, quetiapine, aripiprazole, ziprasidone, iloperidone, lurasidone, paliperidone, brexpiprazole or cariprazine) that is not prescribed as a PRN medication;

Exclusion Criteria:

1. Patients will be excluded if they have had exposure to a total daily dose of MET 1000 mg bid for at least 2 weeks in the past 3 months;
2. Patients will be excluded if they could not tolerate MET during the recommended titration schedule outlined in the protocol;
3. Major neurological or medical illnesses that affect weight gain (e.g., unstable thyroid disease) or require a systemic medication that might impact weight or glucose regulation (e.g., diabetes mellitus [insulin], chronic renal failure [steroids]);
4. Fasting glucose ≥ 126 mg/dL on 2 occasions during screening indicating need for prompt treatment;
5. If lab results are available in the last 6 months, then a serum creatinine ≥1.3 mg/dL on 2 occasions during screening and/or follow-up, indicating potential impairment of renal functioning;
6. Pregnant or breast feeding;
7. Children and caregivers who are unable to complete assessments for any reason;

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1565 (Actual)
Dates: Start 2015-12; Primary Completion 2022-12 (Actual); Study Completion 2023-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P DelBello, MD, MS, Principal Investigator — University of Cincinnati
Locations (29):
- United States (29):
  - The Children's Home of Northern Kentucky, Covington, Kentucky
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - South Oaks, Amityville, New York
  - SUNY Downstate/ Kings County Hospital, Brooklyn, New York
  - Maimonides, Brooklyn, New York
  - NYCCC, Brooklyn, New York
  - Northwell Zucker Long Island Jewish Hospital, Glen Oaks, New York
  - Mount Sinai, New York, New York
  - LIJ Zucker Hillside Hospital, New York, New York
  - Child Center of New York,, Queens, New York
  - NorthShore Child and Family Guidance, Roslyn Heights, New York
  - StonyBrook, Stony Brook, New York
  - Lighthouse Youth Services, Cincinnati, Ohio
  - Central Clinic, Cincinnati, Ohio
  - Children's Home, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Resident Mood Medication Clinic, Cincinnati, Ohio
  - St. Aloysius, Cincinnati, Ohio
  - Talbert House, Cincinnati, Ohio
  - St. Joseph's Orphanage, Cincinnati, Ohio
  - Child Focus, Cincinnati, Ohio
  - NECCO, Cincinnati, Ohio
  - University Hospital Medical Center Cleveland, Cleveland, Ohio
  - Nationwide Children's Hospital Columbus, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - South Community, Dayton, Ohio
  - Butler Behavioral Health Services, Hamilton, Ohio
  - TCN Family Solutions, Xenia, Ohio
  - Seton Family of Hospitals, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DelBello MP, Welge JA, Klein CC, Blom TJ, Fornari V, Higdon C, Sorter MT, Kurtz B, Starr C, Smith A, Huang B, Chen C, Modi AC, Crimmins N, Correll CU; MOBILITY Consortium. Metformin for overweight and obese children and adolescents with bipolar spectrum and related mood disorders treated with second-generation antipsychotics: a randomised, pragmatic trial. Lancet Psychiatry. 2025 Dec;12(12):893-905. doi: 10.1016/S2215-0366(25)00273-1. PMID 41233082
- [Derived] Higdon C, Welge JA, Crimmins NA, Klein CC, Fornari VM, Sorter MT, Blom TJ, Kurtz BP, Correll CU, DelBello MP. Metabolic syndrome in youth with bipolar spectrum disorders treated with second-generation antipsychotics: baseline results from the community-based pragmatic MOBILITY Trial. Eur Child Adolesc Psychiatry. 2025 Sep;34(9):2917-2929. doi: 10.1007/s00787-025-02680-2. Epub 2025 Apr 11. PMID 40214755
- [Derived] Welge JA, Correll CU, Sorter MT, Fornari VM, Blom TJ, Carle AC, Huang B, Klein CC, DelBello MP. Metformin for Overweight and Obese Children With Bipolar Spectrum Disorders Treated With Second-Generation Antipsychotics (MOBILITY): Protocol and Methodological Considerations for a Large Pragmatic Randomized Clinical Trial. JAACAP Open. 2023 Mar 13;1(1):60-73. doi: 10.1016/j.jaacop.2023.03.004. eCollection 2023 Jun. PMID 39554834
- See also: US Centers for Disease Control and Prevention growth charts — https://www.cdc.gov/growthcharts/index.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1633 participants were screened. 68 did not meet criteria. Of the 1565 randomized patients, 228 patients did not have a visit after baseline and 38 patients, in the MET+LIFE group, did not start metformin per protocol by study day 137 post-randomization. These 266 patients were not included in the modified intent-to-treat (ITT) sample and results, giving an ITT sample size of 1299.
Period: Overall Study
Arm/Group | MET and LIFE | Healthy Lifestyle Intervention (LIFE)
Started | 579 | 720
Followed Randomized Treatment (Per-protocol Sample) | 558 | 686
Completed | 360 | 454
Not Completed | 219 | 266
Not completed — Withdrawal by Subject | 12 | 2
Not completed — Lost to Follow-up | 119 | 126
Not completed — Discharged from Clinic Services | 53 | 84
Not completed — Censored (study ended before participant could complete) | 18 | 24
Not completed — Follow-up at non-study site | 8 | 16
Not completed — Moved from area | 9 | 14

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat sample, which includes all randomized patients who had a post-randomization visit and started their randomized intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | MET and LIFE | Healthy Lifestyle Intervention (LIFE) | Total
Number analyzed (Participants) | 579 | 720 | 1299
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.0 (2.8) | 13.8 (2.9) | 13.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273 | 341 | 614
  Male | 306 | 379 | 685
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 96 | 156
  Not Hispanic or Latino | 517 | 624 | 1141
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 11 | 13 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 98 | 124 | 222
  White | 399 | 472 | 871
  More than one race | 50 | 78 | 128
  Unknown or Not Reported | 17 | 29 | 46
BMI Z-Score [Mean (Standard Deviation); unit: Z-score] — Raw body mass index (BMI) is calculated as (weight(kg)/ height(m)2). This raw BMI value is converted to a normalized BMI z-score, adjusted for age and sex using US Centers for Disease Control and Prevention growth charts. A z-score equal to 0 indicates the population mean and larger z-scores are heavier weights and worse outcomes.
  Z-score | 1.90 (0.48) | 1.85 (0.46) | 1.87 (0.47)
Obesity [Count of Participants; unit: Participants] — BMI greater or equal to 95th percentile for age and sex
  Participants | 385 | 474 | 859

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI Z-score From Baseline to Month 6 in ITT Sample
Description: Raw body mass index (BMI) is calculated as (weight(kg)/ height(m)2). This raw BMI value is converted to a normalized BMI z-score, adjusted for age and sex using US Centers for Disease Control and Prevention growth charts. A z-score equal to 0 indicates the population mean and larger z-scores are heavier weights and worse outcomes.
Time Frame: Baseline to Month 6
Population: Modified intention-to-treat (ITT) sample consisting of patients who initiated randomized treatment and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | MET and LIFE | Healthy Lifestyle Intervention (LIFE)
Number analyzed (Participants) | 565 | 687
Z-score | -0.08 (0.29) | 0.00 (0.29)
Statistical Analysis 1: Comparison: MET and LIFE vs Healthy Lifestyle Intervention (LIFE); Test type: Superiority; p < 0.001, ANCOVA — This is a calculated p-value less than 0.001; Mean Difference (Net) = 0.08

2. Primary Outcome: Change in BMI Z-score From Baseline to Month 24 in ITT Sample
Description: as for outcome 1
Time Frame: Baseline to Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | MET and LIFE | Healthy Lifestyle Intervention (LIFE)
Number analyzed (Participants) | 579 | 720
Z-score | -0.19 (1.00) | -0.11 (0.87)
Statistical Analysis 1: Comparison: MET and LIFE vs Healthy Lifestyle Intervention (LIFE); Test type: Superiority; p = 0.044, ANCOVA; Mean Difference (Net) = 0.07

3. Primary Outcome: Change in BMI Z-score From Baseline to Month 6 in Per Protocol Sample
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Per protocol sample consisting of patients who had continuously followed their randomized treatment through month 6
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | MET and LIFE | Healthy Lifestyle Intervention (LIFE)
Number analyzed (Participants) | 547 | 656
Z-score | -0.09 (0.46) | 0.00 (0.42)
Statistical Analysis 1: Comparison: MET and LIFE vs Healthy Lifestyle Intervention (LIFE); Test type: Superiority; p < 0.001, ANCOVA — This is a calculated p-value less than 0.001; Mean Difference (Net) = 0.08

4. Primary Outcome: Change in BMI Z-score From Baseline to Month 24 in Per Protocol Sample
Description: as for outcome 1
Time Frame: Baseline to Month 24
Population: Per protocol sample consisting of patients who had continuously followed their randomized treatment through month 24
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | MET and LIFE | Healthy Lifestyle Intervention (LIFE)
Number analyzed (Participants) | 558 | 686
Z-score | -0.21 (1.11) | -0.12 (1.01)
Statistical Analysis 1: Comparison: MET and LIFE vs Healthy Lifestyle Intervention (LIFE); Test type: Superiority; p = 0.041, ANCOVA; Mean Difference (Net) = 0.09

ADVERSE EVENTS:
Time Frame: 30 months
Description: Other non-serious adverse events are reported for the per protocol sample, consisting of patients who had followed their randomized treatment.
Arm/Group | MET and LIFE | Healthy Lifestyle Intervention (LIFE)
All-Cause Mortality (participants affected / at risk) | 0/579 | 0/720
Serious Adverse Events (participants affected / at risk) | 12/579 | 25/720
Other Adverse Events (participants affected / at risk) | 352/558 | 339/686
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MET and LIFE (N=579) | Healthy Lifestyle Intervention (LIFE) (N=720)
abdominal pain (General disorders) | 5 | 1
refractory headaches (General disorders) | 2 | 0
complications of tonsillectomy (General disorders) | 2 | 2
neck dystonia (General disorders) | 1 | 0
seizures (General disorders) | 1 | 2
hypoglycemia (General disorders) | 1 | 0
pneumonia (General disorders) | 0 | 3
pyelonephritis (General disorders) | 0 | 3
urethral/kidney stone (General disorders) | 0 | 3
infection (General disorders) | 0 | 3
hepatitis (General disorders) | 0 | 1
allergic reaction (General disorders) | 0 | 2
fractures due to motor vehicle accident (General disorders) | 0 | 1
thyroidectomy (General disorders) | 0 | 1
leukemia (General disorders) | 0 | 1
sickle-cell crisis (General disorders) | 0 | 1
Sydenham's Chorea (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MET and LIFE (N=558) | Healthy Lifestyle Intervention (LIFE) (N=686)
Increased Appetite (General disorders) | 56 | 91
Sedation (General disorders) | 20 | 41
Headache (General disorders) | 24 | 31
Somnolence (General disorders) | 14 | 20
Fatigue (General disorders) | 11 | 21
Nausea (Gastrointestinal disorders) | 117 | 69
Diarrhea (Gastrointestinal disorders) | 105 | 40
Vomiting (Gastrointestinal disorders) | 70 | 32
Stomach Cramps (Gastrointestinal disorders) | 110 | 57
Flatulence (Gastrointestinal disorders) | 83 | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT02515773/Prot_SAP_000.pdf